CLINICAL TRIAL: NCT06687902
Title: Added Value of Digital Breast Tomosynthesis in Characterization of Breast Lesions
Brief Title: Value of Digital Breast Tomosynthesis in Breast Lesions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shorouk Salaheldien Ali, M.B.B.Ch, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-15-10---5MS
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Digital Breast Tomosynthesis
MeSH Terms: interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with breast lesions (Experimental)
  Interventions: Diagnostic Test: Digital breast tomosynthesis

INTERVENTIONS:
Diagnostic Test: Digital breast tomosynthesis — In digital breast tomosynthesis (DBT), images are acquired using a specialized X-ray tube that moves in an arc around the breast. This technique captures multiple low-dose images from various angles, typically within a 15° to 60° range. These images are then reconstructed into 1-mm slices to create a 3D representation of the breast, allowing for detailed layer-by-layer evaluation. The number of images acquired varies depending on the size of the breast and the specifications of the equipment but generally ranges from 10 to 25 projections, captured within a few seconds.

SUMMARY:
The aim of the study is to evaluate the added value of digital breast tomosynthesis (DBT) in the characterization of breast lesions.

DETAILED DESCRIPTION:
All patients enrolled in the study will undergo both 2D digital mammography and digital breast tomosynthesis (DBT), using standardized protocols. The DM plus DBT acquisition commonly referred to as "combo" mode , that has shown an improvement in specificity and sensitivity , but at approximately doubling of the radiation dose . This approach will provide a consistent framework for evaluating the diagnostic capabilities of both techniques in characterizing breast masses.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mammographic breast lesions of BIRADS III, IV.
2. Dense breast in patients with complaints (BIRADS 0) which needed further assessment.

Exclusion Criteria:

1. Pregnant females to avoid the hazards of ionizing radiation to the fetus.
2. Patients with known metastatic breast cancer.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
Compare DBT with traditional mammography in terms of diagnostic accuracy, sensitivity, and specificity for detecting and differentiating benign and malignant breast lesions | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
for risk of participant data identification and for privacy concerns